CLINICAL TRIAL: NCT02114684
Title: An Open Label Randomized Controlled Clinical Trial Comparing a 24Week Oral Regimen Containing Moxifloxacin With a 24 Week Standard Drug Regimen for the Treatment of Smear-positive Pulmonary Tuberculosis in Patients Previously Treated for TB
Brief Title: Improving Retreatment Success (IMPRESS)
Acronym: IMPRESS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Responsible Party: Principal Investigator, Dr Nesri Padayatchi, Principle Investigator, Centre for the AIDS Programme of Research in South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CAP 011
Record Dates: First submitted 2014-01-29; First posted 2014-04-15 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Recurrent Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin (Active Comparator): A Moxifloxacin-containing oral regimen of Isoniazid (H), Rifampicin (R), Pyrazinamide (Z), Moxifloxacin (M), substituting Moxifloxacin for Ethambutol, daily for 24 weeks, see information below.
  Intensive phase 7 days a week for 8 weeks Continuation phase - 7 days a week for 16 weeks
  RH(150,75mg), Z (500mg), M (400mg) Dosage and number of tablets dispensed is dependent on participants weight band.
  Interventions: Drug: moxifloxacin
- Ethambutol (Active Comparator): An Ethambutol oral regimen of Isoniazid (H), Rifampicin(R), Pyrazinamide (Z), Ethambutol(E), daily for 24 weeks duration, substituting Ethambutol for Moxifloxacin.
  Intensive phase 7 days a week for 8 weeks Continuation phase - 7 days a week for 16 weeks.See details below.
  (150,75,400,275 mg) RHZE Dosage and number of tablets dispensed is dependent on participants weight band.
  Interventions: Drug: moxifloxacin

INTERVENTIONS:
Drug: moxifloxacin — [isoniazid (H), rifampicin (R), pyrazinamide (Z), moxifloxacin (M)]
  Other Names: AVELON

SUMMARY:
This is an open label randomized controlled clinical trial comparing two regimens for treatment of smear-positive pulmonary TB, among patients previously treated for TB. The primary objective is to determine if a moxifloxacin-containing regimen, substituting moxifloxacin for ethambutol, of 24 weeks duration is superior to a control regimen of 24 weeks duration in improving treatment outcomes in patients with recurrent TB and shortens the duration of TB treatment.

DETAILED DESCRIPTION:
Intervention Arm :12 months (6 months treatment + 12 months post treatment follow up) Control Arm :12 months (6 months treatment + 12 months post treatment follow up) Total sample size is 330.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Previous history of anti-TB chemotherapy
* HIV status: HIV infected and uninfected patients are allowed in the study:
* All patients must agree to HIV testing to confirm HIV status.
* Patients already on ARVs will be allowed in the study provided that the ART regimen is not contraindicated with any of the study agents .
* HIV infected patients at any CD4 count irrespective of ART commencement and duration will be included in the study
* Smear positive or Gene Xpert positive pulmonary tuberculosis
* Rifampicin susceptible as determined by Gene Xpert at screening. Gene Xpert will be used to determine rifampicin resistance, hence the study team will made aware of resistance within 48 hours and prior to study enrolment.
* Karnofsky score greater than 70
* Female candidates of reproductive potential must agree to use two reliable methods of contraception while on study: a barrier method of contraception (condoms or cervical cap) together with another reliable form of contraceptive (condoms with a spermicidal agent, a diaphragm or cervical cap with spermicide, an Intrauterine Device (IUD), or hormone-based contraceptive)
* A negative pregnancy test
* Laboratory parameters done at, or 14 days prior to, screening:

  * Haemoglobin level of at least 7.0 g/dL
  * Serum aspartate transaminase (AST) and alanine transaminase (ALT) activity less than 3 times the upper limit of normal
  * Serum total bilirubin level less than 2.5 times upper limit of normal
  * Creatinine clearance (CrCl) level greater than 60 mls/min
  * Platelet count of at least 50 x109cells/L
  * Serum potassium greater than 3.0 mmol/L

Exclusion Criteria:

* Patients on a Nevirapine (NVP)-containing ART regimen at screening
* Pregnant or breastfeeding
* Received an antibiotic active against M. tuberculosis in the last 14 days (e.g. fluoroquinolones, macrolides, standard anti-tuberculosis drugs).
* Patients with known M. tuberculosis resistance to any of the study drugs at screening
* History of prolonged QT syndrome or current or planned therapy with quinidine, procainamide, amiodarone, sotalol, or ziprasidone during the intensive phase of tuberculosis treatment.
* Known allergies or intolerance to any of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nesri Padayatchi, MBChB, MSc, Principal Investigator — Centre for the AIDS Programme of Research in South Africa; Kogieleum Naidoo, MBChB, Study Director — Centre for the AIDS Programme of Research in South Africa
Locations (1):
- CAPRISA eThekwini Clinical Research Site (eCRS), Durban, KwaZulu-Natal, South Africa

REFERENCES:
- [Derived] Rambaran S, Maseko TG, Lewis L, Hassan-Moosa R, Archary D, Ngcapu S, Garrett N, McKinnon LR, Padayatchi N, Naidoo K, Sivro A. Blood monocyte and dendritic cell profiles among people living with HIV with Mycobacterium tuberculosis co-infection. BMC Immunol. 2023 Jul 21;24(1):21. doi: 10.1186/s12865-023-00558-z. PMID 37480005
- [Derived] Perumal R, Padayatchi N, Yende-Zuma N, Naidoo A, Govender D, Naidoo K. A Moxifloxacin-based Regimen for the Treatment of Recurrent, Drug-sensitive Pulmonary Tuberculosis: An Open-label, Randomized, Controlled Trial. Clin Infect Dis. 2020 Jan 1;70(1):90-98. doi: 10.1093/cid/ciz152. PMID 30809633
- [Derived] Naidoo A, Chirehwa M, Ramsuran V, McIlleron H, Naidoo K, Yende-Zuma N, Singh R, Ncgapu S, Adamson J, Govender K, Denti P, Padayatchi N. Effects of genetic variability on rifampicin and isoniazid pharmacokinetics in South African patients with recurrent tuberculosis. Pharmacogenomics. 2019 Mar;20(4):225-240. doi: 10.2217/pgs-2018-0166. Epub 2019 Feb 15. PMID 30767706

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One individual in the control arm was terminated one month after enrollment owing to discovery of pre-existing violation of entry criteria. The individual was excluded from all statistical analyses.
Groups:
- Moxifloxacin: A Moxifloxacin-containing oral regimen of Isoniazid (H), Rifampicin (R), Pyrazinamide (Z), Moxifloxacin (M), substituting Moxifloxacin for Ethambutol.
  The intervention arm substituted moxifloxacin for ethambutol (moxifloxacin group), and consisted of daily doses of moxifloxacin, rifampicin, isoniazid and pyrazinamide for 8 weeks, followed by daily doses of moxifloxacin, rifampicin and isoniazid for 16 weeks.
  Participants in the moxifloxacin arm received daily 400 mg of moxifloxacin (Avelox®, Bayer Healthcare), weight-based rifampicin at 450 or 600 mg, and 225 or 300 mg of isoniazid, for participants 38-54 and ≥55 kg, respectively, during the 2-month intensive phase and 4-month continuation phase of TB treatment. During the intensive phase of treatment, pyrazinamide was used at 1500 and 2000mg in participants between 38-54 and ≥55 kg, respectively.
- Control: An Ethambutol oral regimen of Isoniazid (H), Rifampicin(R), Pyrazinamide (Z), Ethambutol(E), substituting Ethambutol for Moxifloxacin.
  Daily doses of rifampicin, isoniazid, pyrazinamide and ethambutol for 8 weeks (intensive phase), followed by daily doses of rifampicin and isoniazid for 16 weeks (Continuation phase).
  During the first two months (intensive phase) of treatment, participants in the control arm received the following weight-based doses by fixed dose combination tablets: Participants who were 38 - 54kg received rifampicin 450mg, isoniazid 225mg, pyrazinamide 1200mg, ethambutol 825mg; participants who were 54 - 70kg received rifampicin 600mg, isoniazid 300mg, pyrazinamide 1600mg, ethambutol 1100mg; participants who were > 70 kg received rifampicin 750mg, isoniazid 375mg, pyrazinamide 2000mg, ethambutol 1375mg. During the subsequent four months (continuation phase), participants continued on the same weight-based doses of rifampicin and isoniazid.
Period: Overall Study
Arm/Group | Moxifloxacin | Control
Started | 98 | 98
Completed | 86 | 88
Not Completed | 12 | 10
Not completed — Death | 6 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Relocation | 3 | 1
Not completed — Rifampicin resistant on culture | 0 | 1
Not completed — Patient Incarcerated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin | Control | Total
Number analyzed (Participants) | 98 | 98 | 196
Age, Customized [Count of Participants; unit: Participants]
  <25 years | 7 | 14 | 21
  =>25 and <35 years | 37 | 35 | 72
  =>35 and <=45 years | 35 | 32 | 67
  >45 years | 19 | 17 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 35 | 59
  Male | 74 | 63 | 137
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 96 | 98 | 194
  White | 1 | 0 | 1
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 98 | 98 | 196

OUTCOME MEASURES:

1. Primary Outcome: Sputum Culture Conversion Rates at Week 8 and Month 6 Post Tuberculosis Treatment Initiation
Description: The proportion of patients with negative sputum cultures at the end of the intensive phase (8 weeks) and the proportion of patients with negative sputum cultures at 6 months were compared between the two study arms. All participants with sputum culture results at week 8 and month 6 were included in the analysis.
Time Frame: 24 weeks
Population: Nine participants had missing data at week 8: 4 missed visits, 3 terminated before week 8 and 2 had MOTT cultured. Fourteen had missing data at month 6: 7 were terminated before month 6 and 7 missed their visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Moxifloxacin | Control
Number analyzed (Participants) | 98 | 98
Participants
  culture negative at 8 weeks: number analyzed (Participants) | 94 | 93
  culture negative at 8 weeks | 78 | 73
  culture negative at 6 months: number analyzed (Participants) | 88 | 94
  culture negative at 6 months | 84 | 92
Statistical Analysis 1: Comparison: Moxifloxacin vs Control; comparison of culture negative results at week 8; Test type: Superiority; p = 0.46, Fisher Exact
Statistical Analysis 2: Comparison: Moxifloxacin vs Control; comparison of culture negative results at month 6; Test type: Superiority; p = 0.43, Fisher Exact

2. Secondary Outcome: Time to Culture-conversion of the Moxifloxacin Regimen and the Ethambutol Regimen
Description: To determine the time to culture-conversion of the moxifloxacin regimen and the ethambutol regimen.
Time Frame: Up to 2 years
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Moxifloxacin | Control
Number analyzed (Participants) | 98 | 98
weeks | 6.0 [4.0 to 8.3] | 7.9 [4.0 to 11.4]
Statistical Analysis 1: Comparison: Moxifloxacin vs Control; Test type: Superiority; p = 0.018, Gehan-Breslow-Wilcoxon test

3. Secondary Outcome: Proportion of Patients With Any Grade 3 or 4 Adverse Reactions in the Two Study Arms
Description: To compare the proportion of patients with any Grade 3 or 4 adverse reactions in the two study arms. Outcome measured in terms of number of participants with at least one grade 3 or 4 events, and not in number of events.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Moxifloxacin | Control
Number analyzed (Participants) | 98 | 98
Participants | 43 | 25
Statistical Analysis 1: Comparison: Moxifloxacin vs Control; Test type: Superiority; p = 0.011, Fisher Exact

4. Secondary Outcome: Number of Participants With Adverse Events and 8-week Culture Conversion Rates Among HIV-infected Patients vs. HIV-uninfected Patients
Description: To compare adverse events and 8-week culture conversion rates among HIV-infected patients vs. HIV-uninfected patients. The proportion of participants with at least one grade 3 or 4 adverse event was measured.
Time Frame: up to 2 years for adverse events and 8 weeks for culture conversion rates
Population: 9 participants had missing data at 8 weeks: 4 missed visits, 3 terminated before week 8, and 2 had MOTT cultured
Measure: Count of Participants; unit: Participants
Groups:
- HIV Positive, Moxifloxacin: HIV negative participants based on HIV status at study enrollment, who were assigned to the Moxifloxacin group
- HIV Positive, Control: HIV positive participants based on HIV status at study enrollment, who were assigned to the control group
- HIV Negative, Moxifloxacin: HIV negative participants based on HIV status at study enrollment, who were assigned to the Moxifloxacin arm
- HIV Negative, Control: HIV negative participants based on HIV status at study enrollment, who were assigned to the control group
Arm/Group | HIV Positive, Moxifloxacin | HIV Positive, Control | HIV Negative, Moxifloxacin | HIV Negative, Control
Number analyzed (Participants) | 70 | 68 | 28 | 30
Participants
  participants with grade 3/4 adverse events | 30 | 19 | 13 | 6
  participants culture negative at 8 weeks: number analyzed (Participants) | 67 | 64 | 27 | 29
  participants culture negative at 8 weeks | 57 | 51 | 21 | 22
Statistical Analysis 1: Comparison: HIV Positive, Moxifloxacin vs HIV Positive, Control vs HIV Negative, Moxifloxacin vs HIV Negative, Control; Comparison of the number of adverse events in the two arms, controlling for HIV status; Test type: Superiority; p = 0.01, Mantel Haenszel — There are significantly more adverse events in the active arm
Statistical Analysis 2: Comparison: HIV Positive, Moxifloxacin vs HIV Positive, Control vs HIV Negative, Moxifloxacin vs HIV Negative, Control; Comparison of the 8-week culture conversion rates in the two arms, controlling for HIV status; Test type: Superiority; p = 0.45, Mantel Haenszel

5. Secondary Outcome: Proportion of Patients With Unfavourable Outcomes or Tuberculosis Recurrence in the Moxifloxacin and Control Arm.
Description: A patient was defined as having an unfavourable outcome if he/she was not cured at the end of treatment or did not successfully complete treatment. Recurrence after completion of treatment was defined as two positive cultures within a period of four months without an intervening negative culture.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Moxifloxacin | Control
Number analyzed (Participants) | 98 | 98
Participants | 13 | 6
Statistical Analysis 1: Comparison: Moxifloxacin vs Control; Test type: Superiority; p = 0.15, Fisher Exact

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Moxifloxacin | Control
All-Cause Mortality (participants affected / at risk) | 6/98 | 4/98
Serious Adverse Events (participants affected / at risk) | 27/98 | 12/98
Other Adverse Events (participants affected / at risk) | 30/98 | 19/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxifloxacin (N=98) | Control (N=98)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 4 (4)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site paraesthesia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Treatment failure (General disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound sepsis (Infections and infestations) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Epidemic vomiting syndrome (Infections and infestations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Neurological examination abnormal (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Blood osmolarity decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bach's flower remedy (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxifloxacin (N=98) | Control (N=98)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 6 (7) | 2 (2)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sputum purulent (Infections and infestations) | 0 (0) | 1 (1)
Bone tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Extrapulmonary tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 5 (5) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Female reproductive tract carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (3)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-05-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT02114684/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT02114684/SAP_001.pdf